CLINICAL TRIAL: NCT01679405
Title: Open-label, Uncontrolled, Multicenter Phase I/Ib Trial to Investigate Safety and Efficacy of BIBW 2992 and Standard Gemcitabine/Cisplatin in Chemo-naïve Patients With Advanced Biliary Tract Adenocarcinoma
Brief Title: BIBW 2992 as add-on to Gem/Cis in Advanced Biliary Tract Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: No sufficient clinical or molecular signals for efficacy were observed.
Sponsor: Johannes Gutenberg University Mainz (Other)
Responsible Party: Principal Investigator, PD Dr Markus Möhler, Principal Investigator, Johannes Gutenberg University Mainz
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BIBW 2992
Record Dates: First submitted 2012-08-17; First posted 2012-09-06 (Estimated); Results first posted 2019-01-22 (Actual); Last update posted 2019-09-06 (Actual); Status verified 2019-08

CONDITIONS: Metastatic Disease
Keywords: metastatic biliary tract cancer
MeSH Terms: conditions — Neoplasm Metastasis; Biliary Tract Neoplasms | interventions — Afatinib; Gemcitabine; Cisplatin

STUDY DESIGN:
Intervention Model Description: For Part A of the study a standard 3+3 design was used. The recruitment was carried out in cohorts. Subjects were not allowed to participate in both cohorts. If the maximum tolerated dose was found there should be additional patients recruited to confirm the maximum tolerated dose (part B)
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dose level 1 (Part A) (Experimental): 30 mg BIBW 2992, Gemcitabin (1.000 mg/m² BSA i.v.)/Cisplatin (25 mg/m² BSA i.v.)
  Interventions: Drug: BIBW 2992
- Dose level -1 (Part A) (Experimental): 30 mg BIBW 2992, Gemcitabin (800 mg/m² BSA i.v.)/Cisplatin (20 mg/m² BSA i.v.)
  Interventions: Drug: BIBW 2992

INTERVENTIONS:
Drug: BIBW 2992 — once daily per os
  Other Names: Gemcitabine and Cisplatin

SUMMARY:
An open-label, uncontrolled, multicenter phase I/Ib trial to investigate safety and efficacy of BIBW 2992 added to the standard therapy of Gemcitabine/Cisplatin in chemo-naïve patients with advanced and/or metastatic adenocarcinoma of the biliary tract

DETAILED DESCRIPTION:
The primary objective is safety and toxicity, including maximum tolerated dose, of BIBW 2992 when given as add-on therapy to Gem/Cis.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients aged ≥ 18 years
* Signed and dated written informed consent,
* Histologically confirmed adenocarcinoma of the gallbladder or intrahepatic bile ducts or extrahepatic bile ducts (metastasized) or histologically proven hepatic metastases of an earlier resected and histologically proven biliary tract cancer or a Klatskin tumour (hilar cholangiocarcinoma)

  * with pain and biliary obstruction controlled
  * adequate biliary drainage, no uncontrolled infection
  * ECOG Performance Status of 0-1
  * LFTs: bilirubin (total) ≤ 1.5 x ULN, ALT/ AST/ alkaline phosphatase ≤ 3 2.5 x ULN (≤ 5 x ULN if liver metastases are present)
  * No prior systemic treatment i) previous adjuvant chemotherapy is allowed (completed ≥ 6 months if containing Gemcitabine or platinum salts); ii) previous irradiation (external radiotherapy, brachytherapy, chemoembolization) and PDT are allowed, provided that there is still at least one unidimensionally measurable target lesion in an untreated area
* Resolution of all side effects of prior surgical procedures to CTCAE grade ≤ 1 (except for the laboratory values specified below)
* At least 4 weeks from any major surgery (at first dose of study drug)
* Life expectancy of at least 12 weeks.
* Cardiac left ventricular function with resting ejection fraction (LVEF) ≥ 50%
* Adequate bone marrow, liver and renal function as assessed by the following laboratory requirements to be conducted within 7 days prior to start of therapy:

  * Haemoglobin > 10.0 g/dl (=6.2 mmol/l), blood transfusion is allowed
  * Absolute neutrophil count (ANC) > 1,500/mm3 (=1.5x 109/L)
  * Platelet count ≥ 100,000/μl (=100x 109/L)
  * Total bilirubin ≤ 1.5 times the upper limit of normal
  * ALT and AST ≤ 2.5 x institutional upper limit of normal (in case of liver metastases: ALT and AST ≤ 5 x institutional upper limit of normal)
  * Prothrombin rate > 60% or INR < 1.5

Main exclusion criteria

* Large surgery (except diagnostic biopsy) or smaller surgical procedures, external radiotherapy, brachytherapy, or PDT within 30 days prior to start of treatment.
* Other tumor type than adenocarcinoma (e.g. leiomyosarcoma, lymphoma) or a second cancer except in patients with squamous or basal cell carcinoma of the skin or carcinoma in situ of the cervix which has been effectively treated.
* History of acute cardiac disease: congestive heart failure > NYHA class 2; active CAD (MI more than 6 months prior to study entry is allowed);
* Patients on immunosuppressant therapy or with known HIV infection
* Active clinically serious infections (> grade 2 NCI-CTC version 3.0)
* History of organ allograft
* Pregnant or breast-feeding patients.
* Substance abuse, medical, psychological or social conditions that may interfere with the patient's participation
* Any condition that is unstable or could jeopardize the safety of the patient and their compliance in the study
* Gastrointestinal (GI) tract disease resulting in an inability to take oral medication or a requirement for IV alimentation, prior surgical procedures affecting absorption, or active peptic ulcer disease
* History of pre-existing interstitial lung disease (ILD)
* Patients with untreated or symptomatic brain metastases.
* Persistent Grade 2 or greater neurotoxicity / neuropathy from any cause

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2012-08; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Markus Moehler, Prof. Dr. med., Principal Investigator — University Medical Center of the Johannes Gutenberg-University Mainz
Locations (1):
- I. Medizinische Klinik und Poliklinik der Universitätsmedizin, Mainz, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Moehler M, Maderer A, Ehrlich A, Foerster F, Schad A, Nickolay T, Ruckes C, Weinmann A, Sivanathan V, Marquardt JU, Galle PR, Woerns M, Thomaidis T. Safety and efficacy of afatinib as add-on to standard therapy of gemcitabine/cisplatin in chemotherapy-naive patients with advanced biliary tract cancer: an open-label, phase I trial with an extensive biomarker program. BMC Cancer. 2019 Jan 11;19(1):55. doi: 10.1186/s12885-018-5223-7. PMID 30634942

RESULTS

PARTICIPANT FLOW:
Groups:
- Dose Level 1: 30 mg BIBW 2992, Gemcitabine (1.000 mg/m² BSA i.v.)/Cisplatin (25 mg/m² BSA i.v.)
- Dose Level -1: 30 mg BIBW 2992, Gemcitabine (800 mg/m² BSA i.v.)/Cisplatin (20 mg/m² BSA i.v.)
Period: Overall Study
Arm/Group | Dose Level 1 | Dose Level -1
Started | 3 | 6
Completed | 1 | 1
Not Completed | 2 | 5
Not completed — Death | 2 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dose Level 1 | Dose Level -1 | Total
Number analyzed (Participants) | 3 | 6 | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.00 (21.63) | 60.17 (7.31) | 60.78 (12.30)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 3 | 4
  Male | 2 | 3 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 3 | 6 | 9
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Germany | 3 | 6 | 9

OUTCOME MEASURES:

1. Primary Outcome: Number of Adverse Events
Description: In part A the maximum tolerated dose (MTD) of BIBW 2992 administered continuously to the standard therapy of Gemcitabine / Cisplatin (Gem/Cis) (administered together on day 1 and 8 of a three-week cycle) will be evaluated in a 2 step dose escalation.
  Safety and toxicity will be evaluated as described and considered primary for part B of the study.
Time Frame: Treatment period: up to eight cycles (maximum 8 months). 12 months follow-up period.
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Level 1 | Dose Level -1
Number analyzed (Participants) | 3 | 6
Participants | 2 | 1

2. Secondary Outcome: Time to Progress (TTP)
Description: Median time to progress (according to RECIST 1.1 criteria) including the 95% confidence intervals were determined using Kaplan-Meier estimates. Time from start of treatment to first documentation of objective tumour progression. Deaths were censored at the time of death.
Time Frame: Treatment period: up to eight cycles (maximum 8 months). 12 months follow-up period.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Dose Level 1 | Dose Level -1
Number analyzed (Participants) | 3 | 6
days | 159 [134 to 184] | NA [49 to NA] — Median and upper confidence limit could not be calculated, because of too few events.

3. Secondary Outcome: Overall Survival (OS)
Description: Median overall survival time including the 95% confidence interval were determined using Kaplan-Meier estimates.
Time Frame: Time from start of treatment to death due to any cause. Time to last observation will be used if a patient has not died and OS for the patient will be considered censored. Estimated time period: up to 76 weeks
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Dose Level 1 | Dose Level -1
Number analyzed (Participants) | 3 | 6
days | 163 [79 to NA] — Upper confidence limit could not be calculated, because of too few events. | 260 [75 to NA] — Upper confidence limit could not be calculated, because of too few events.

4. Secondary Outcome: Objective Response Rate
Description: Response was assessed by means of RECIST 1.1 criteria for target lesions, non-target lesions and the appearance of new lesions. Objective response was defined as the CR, PR or SD at end of treatment
Time Frame: Treatment period: up to eight cycles (maximum 8 months).
Population: For one patient, there was no CT assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Level 1 | Dose Level -1
Number analyzed (Participants) | 2 | 6
Participants | 0 | 0

5. Secondary Outcome: Tumor Control Rate
Description: Tumor control rate is defined as the best tumour response (confirmed partial or complete response, stable disease) that is achieved until end of treatment according to Recist 1.1.
Time Frame: Treatment period: up to eight cycles (maximum 8 months).
Population: For one patient there was no CT assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Level 1 | Dose Level -1
Number analyzed (Participants) | 2 | 6
Participants | 0 | 4

ADVERSE EVENTS:
Arm/Group | Dose Level 1 | Dose Level -1
All-Cause Mortality (participants affected / at risk) | 2/3 | 5/6
Serious Adverse Events (participants affected / at risk) | 2/3 | 5/6
Other Adverse Events (participants affected / at risk) | 3/3 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose Level 1 (N=3) | Dose Level -1 (N=6)
Progression of disease (fatal) (General disorders) | 1 (1) | 0 (0)
thrombocytopenia, anaemia, hypokaliemia (Investigations) | 1 (1) | 0 (0)
worsening of pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
liver failure (Hepatobiliary disorders) | 0 (0) | 1 (1)
diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1)
diarrhea, hypokaliemia (Gastrointestinal disorders) | 0 (0) | 1 (1)
sepsis, chronic kidney disease (worsening), platelet count decreased, worsening of anemia, diarrhea (Infections and infestations) | 0 (0) | 1 (1)
Infection unknown origin, platelet count decreased (Infections and infestations) | 0 (0) | 1 (1)
"infection unknown origin, worsening of chronic kidney disease, platelet count decreased, leukocytop (Infections and infestations) | 0 (0) | 1 (1)
Biliary tract infection (Infections and infestations) | 0 (0) | 1 (1)
infection, unknown origin, pulmonary embolism both sides, deep vein thrombosis both leg (Infections and infestations) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose Level 1 (N=3) | Dose Level -1 (N=6)
fatigue (General disorders) | 3 (11) | 6 (19)
nausea (Gastrointestinal disorders) | 3 (5) | 5 (9)
diarrhoea (Gastrointestinal disorders) | 2 (4) | 5 (25)
rash (Skin and subcutaneous tissue disorders) | 3 (7) | 4 (10)
stomatitis (Gastrointestinal disorders) | 3 (6) | 4 (8)
anemia (Blood and lymphatic system disorders) | 3 (7) | 4 (8)
weight loss (Investigations) | 1 (2) | 6 (9)
epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 2 (2)
neutropenia (Investigations) | 2 (11) | 3 (9)
thrombocytopenia (Investigations) | 3 (17) | 3 (20)
hypokalemia (Metabolism and nutrition disorders) | 2 (4) | 3 (6)
paresthesia (Nervous system disorders) | 1 (1) | 4 (9)
paronychia (Infections and infestations) | 1 (1) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes